CLINICAL TRIAL: NCT05234502
Title: Effects of Ketogenic Diet on Metabolism and Polyneuropathy in Overweight and Obese Women With Breast Cancer
Brief Title: Effects of Ketogenic Diet in Overweight and Obese Women With Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Mehmet Artac, Proffessor Doctor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Ketogenic Diet
Record Dates: First submitted 2022-01-13; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer Female
Keywords: neoadjuvant chemotherapy; ketogenic diet; polyneuropathy
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Ketogenic diet) (Experimental): Group-1 will be given an adequate and balanced healthy diet program during the standard neoadjuvant treatment (12 weeks) with an anthracycline. And simultaneously with standard neoadjuvant therapy containing taxane (12 weeks), KD will be planned for Group-1
  Interventions: Other: Adequate and balanced healthy diet program (CHO: 45-60%, protein:10-20%, fat:20-35%); Other: Ketogenic diet program (CHO: 6%, protein:19%, fat:75%)
- Group-2 (Adequate and balanced healthy diet) (Other): Group-2 will be given an adequate and balanced healthy diet program during the standard neoadjuvant treatment (12 weeks) with anthracycline and taxane (12 weeks).
  Interventions: Other: Adequate and balanced healthy diet program (CHO: 45-60%, protein:10-20%, fat:20-35%)

INTERVENTIONS:
Other: Adequate and balanced healthy diet program (CHO: 45-60%, protein:10-20%, fat:20-35%) — In calculating the estimated basal metabolic rate of individuals, Mifflin-St. The Jeor Equation will be used.BMR will be multiplied by the physical activity factor of the individual and 500*700 kcal will be subtracted from the found value and the total daily energy requirement will be obtained.
Other: Ketogenic diet program (CHO: 6%, protein:19%, fat:75%) — A ketogenic diet will be applied to Group 1 for 12 weeks simultaneously with taxane treatment.
  Arms: Group-1 (Ketogenic diet)

SUMMARY:
Breast cancer is the most common cancer type among women in Turkey and the world. Chemotherapy, surgery, radiotherapy, immunotherapy and hormone therapy are used in the treatment. Nutrition is one of the important factors affects cancer treatment. In recent years, there has been an increase in the number of clinical studies on the ketogenic diet (KD) in different types of cancer. In the literature, it has been shown the KD applied with chemotherapy improves the quality of life and decreases the body weight and tumour size in women with breast cancer. However, there is no comprehensive study evaluating the effect of KD on chemotherapy-induced sensory and motor neuropathy and survival in breast cancer patients. In this project, the KD will be planned for overweight and obese women diagnosed with breast cancer who will be treated with neoadjuvant chemotherapy. Tumour size, nutritional status, biochemical findings, anthropometric measurements, quality of life, sensory and motor polyneuropathy and survival will be evaluated. Fifty-six women with breast cancer who comply with the study criteria and are willing to participate in the study will be given an adequate and balanced healthy diet program during the standard neoadjuvant treatment (12 weeks) with anthracycline. After the interim evaluation, individuals will be randomly divided into two groups. Simultaneously with standard neoadjuvant therapy containing taxane (12 weeks), KD will be planned for the first group and the second group will continue on the adequate and balanced healthy diet program. After neoadjuvant therapy, the effects of diets on prognosis and other factors (nutritional status, biochemical findings, anthropometric measurements, quality of life, sensory and motor polyneuropathy, and survival) will be compared. In this study, unlike other studies, the first data on the effect of KD on chemotherapy-induced polyneuropathy and pathological response in women with breast cancer will be obtained. In this respect, it has the potential for nutritional practices in clinical oncology. The KD could improve body composition and the complications related to obesity and decrease polyneuropathy. Therefore, drug-using and application to the hospital could decrease. The results of the project will contribute to the improvement of the health and the quality of life of women, who are the most important element of society and the family.

DETAILED DESCRIPTION:
The study was designed as a randomized prospective study.

The Location of the Research: The research will be carried out in Konya Necmettin Erbakan University Meram Faculty of Medicine, Departments of General Surgery, Medical Oncology, and Medical Biochemistry. Ethics committee approval was obtained from the Ethics Committee of Necmettin Erbakan University, (Date:03.09.2021, Number:2021/3378). And the official approval was obtained from the Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician to conduct the study.

The Sample Size of the Study: The study will include overweight and obese female individuals aged 19-64 who volunteered to participate in the study, diagnosed with breast cancer, who applied to Necmettin Erbakan University Meram Faculty of Medicine, Department of General Surgery and planned to receive neoadjuvant treatment in the Department of Medical Oncology. Since the ketogenic diet provides a decrease in body weight and an improvement in body composition, it was decided to include overweight and obese women. Neoadjuvant chemotherapy containing anthracycline and taxane is applied as standard to breast cancer patients in the Department of Medical Oncology of Meram Faculty of Medicine. After neoadjuvant therapy containing anthracyclines, patients will be randomly divided into two groups. A ketogenic diet will be applied to the first group (Group 1), and an adequate and balanced healthy nutrition program will be applied to the second group (Group 2).

The sample size of the study: Considering that the number of samples in Group 1 and Group 2 would be equal, it was determined that both groups should consist of at least 28 individuals with an error margin of d =3, α = 0.05, and a power of 0.90 power and 15% drop rate. In this study, all of the patients participating in the research will be informed in detail and informed consent forms will be obtained from all participants.

Statistical analysis: The data will be assessed using the SPSS 26 statistical software package. Mean, standard deviation, minimum and maximum values of the quantitative data will be calculated, and the number and percentage tables of the qualitative data will be created. In the comparison of quantitative data of Group 1 and 2, the Student t-test will be used for the normal distribution, and the Mann-Whitney U test will be used for the non-normal distribution. The chi-squared test will be used to evaluate qualitative data.

In the comparison of quantitative data of the groups during follow-up one-way ANOVA will be used for the normal distribution, and the Friedman test will be used for the non-normal distribution

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer for the first time,
* Planned to receive neoadjuvant treatment,
* Being overweight (BMI: 25-29.9 kg/m2) or obese (BMI: ≥30 kg/m2),
* Karnofsky Performance Score ≥ 70

Exclusion Criteria:

* Ketogenic diet history,
* Diagnosed with moderate/severe neurological and/or cognitive impairment
* Diagnosed with kidney, liver, and gall bladder disease/coronary artery disease
* Diagnosed with type 1 diabetes,
* Diagnosed with type 2 diabetes using oral antidiabetic or insulin,
* Diagnosed with eating behavior disorder (anorexia nervosa, bulimia nervosa, binge eating disorder),
* Using weight loss medication,
* Karnofsky Performance Score < 70,
* Pregnant
* Breastfeeding individuals

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Breast cancer occurs almost entirely in females.
Enrollment: 56 (Estimated)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Polyneuropathy | 6 months (before and after neoadjuvant therapy)
  Chemotherapy-induced polyneuropathy will be assessed through EORTC QLQ-CIPN20.
Polyneuropathy-severity of symptoms | 6 months (before and after neoadjuvant therapy)
  Severity of symptoms of polyneuropathy will be assessed through National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)
Tumor size | 6 months (before and after neoadjuvant therapy)
  Before and after neoadjuvant therapy, routine radiological imaging report will be evaluated.
Quality of life score-(European Cancer Research and Treatment Organization Quality of Life Scale - Cancer 30 (EORTC QLQ-C30) | 6 months (before and after neoadjuvant therapy)
  The quality of life of women with breast cancer is evaluated with the European Cancer Research and Treatment Organization Quality of Life Scale - Cancer 30 (EORTC QLQ-C30). It consists of 30 items to assess physical, role, emotional, cognitive and social functioning, global health status or qualitiy of life scales, fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties.
Quality of life score-Case group (the European Cancer Research and Treatment Organization Breast Cancer-Specific Quality of Life Scale | 6 months (before and after neoadjuvant therapy)
  The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss.
5-year survival rate | 5 years after neoadjuvant therapy
  After neoadjuvant therapy survival rates will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Burçin ALKAN, MSc, Principal Investigator — Necmettin Erbakan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Cancer Institute. 2017.
- [Background] Postma TJ, Aaronson NK, Heimans JJ, Muller MJ, Hildebrand JG, Delattre JY, Hoang-Xuan K, Lanteri-Minet M, Grant R, Huddart R, Moynihan C, Maher J, Lucey R; EORTC Quality of Life Group. The development of an EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy: the QLQ-CIPN20. Eur J Cancer. 2005 May;41(8):1135-9. doi: 10.1016/j.ejca.2005.02.012. Epub 2005 Apr 14. PMID 15911236
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Khodabakhshi A, Akbari ME, Mirzaei HR, Mehrad-Majd H, Kalamian M, Davoodi SH. Feasibility, Safety, and Beneficial Effects of MCT-Based Ketogenic Diet for Breast Cancer Treatment: A Randomized Controlled Trial Study. Nutr Cancer. 2020;72(4):627-634. doi: 10.1080/01635581.2019.1650942. Epub 2019 Sep 9. PMID 31496287
- [Background] Khodabakhshi A, Akbari ME, Mirzaei HR, Seyfried TN, Kalamian M, Davoodi SH. Effects of Ketogenic metabolic therapy on patients with breast cancer: A randomized controlled clinical trial. Clin Nutr. 2021 Mar;40(3):751-758. doi: 10.1016/j.clnu.2020.06.028. Epub 2020 Jul 3. PMID 32703721
- [Background] Khodabakhshi A, Seyfried TN, Kalamian M, Beheshti M, Davoodi SH. Does a ketogenic diet have beneficial effects on quality of life, physical activity or biomarkers in patients with breast cancer: a randomized controlled clinical trial. Nutr J. 2020 Aug 22;19(1):87. doi: 10.1186/s12937-020-00596-y. PMID 32828130
- See also: Sample Size Calculator — https://riskcalc.org/samplesize